CLINICAL TRIAL: NCT05299307
Title: The Impact of Covid-19 Vaccination on the Reproductive and Sexual Function in Sample of Male Egyptian Population
Brief Title: Effect of Covid-19 Vaccination on Male
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed el mahdy abdelmotaleb, Assistant lecturer, Assiut University
Other Study IDs: Effect of Covid-19 Vaccination
Record Dates: First submitted 2022-03-27; First posted 2022-03-29 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Semen Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: semen analysis and hormonal proflie — measure total prolactin and total testosterone and semen

SUMMARY:
we will assess the effect ofcovid19 vaccination on the reproductive and sexual function of the Male Egyptian

DETAILED DESCRIPTION:
Coronaviruses are a group of RNA viruses that primarily affect the respiratory system and cause the common cold, fever, and coughs in mammals and birds. However, in some cases, coronaviruses are associated with more serious and lethal conditions, such as pneumonia, bronchitis, and severe acute respiratory syndrome .

Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) originating from Wuhan, China, led to a global health crisis. SARS-CoV-2 had infected more than 450 million people, resulting in more than 6.6 million deaths. The World Health Organization (WHO) declared coronavirus disease 2019 (COVID-19), the infectious disease caused by SARS-CoV-2, a pandemic, and many states enacted strict rules, such as border closures, transportation restrictions, and quarantine.

Quality and satisfying sexual life have a positive effect on the social and daily relationships as well as on the intimate life of many individuals. The WHO summarizes the definition of sexual health as the physical, emotional, mental, and social well-being of an individual. On the other hand, sexual dysfunction can be described as any condition preventing the individual from being satisfied by the sexual activity at any stage of the sexual relationship.

The renin-angiotensin system (RAS), also ACE 2 and TMPRSS2 play an important role in the cellular entry for SARS-CoV-2. Because the male genital system presents high ACE 2 expression, the importance of this pathway increases in COVID-19 cases. As the COVID-19 pandemic has affected the male genital system in direct or indirect ways and showed a negative impact on male reproduction Ozer Baran and Aykut Aykac et al reported that the fear of infection and transmission of the disease to the partner that occurs during the Covid-19 pandemic manifests itself in the form of a decrease in the frequency and quality of sexual intercourse.

A COVID 19 vaccine is a biotechnology product intended to provide acquired immunity against corona virus disease 2019 (COVID 19) As of 1st June 2020, there were 124 candidate vaccines that were being developed for the prophylaxis of COVID-19. Of these, 10 vaccine candidates had entered phase1, combined phase 1/2 or phase 2 human clinical trials in adults

ELIGIBILITY:
Inclusion Criteria:

* Male patients receive covid 19 vaccinations. Age from 20 to 55 years

Exclusion Criteria:

* Patients complaining of ED or any sexual dysfunction before Vaccination.

  * Patients with history of male infertility before Vaccination.
  * Patients who have pyschological disorders or any other systemicdiseases

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We shall also compare the sexual function of men as well as the reproductive function of men before and after covid 19 vaccination receiving two doses .We shall also compare the sexual function of men as well as the reproductive function of men after covid 19 vaccination receiving two doses and after receiving 3 doses(booster dose).
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Effect of Covid19 Vaccination on the reproductive and sexual function in a sample of Egyptian population | Baseline
  Analysis the effect of the vaccination on the semen parameters and sexual function

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikari SP, Meng S, Wu YJ, Mao YP, Ye RX, Wang QZ, Sun C, Sylvia S, Rozelle S, Raat H, Zhou H. Epidemiology, causes, clinical manifestation and diagnosis, prevention and control of coronavirus disease (COVID-19) during the early outbreak period: a scoping review. Infect Dis Poverty. 2020 Mar 17;9(1):29. doi: 10.1186/s40249-020-00646-x. PMID 32183901
- [Background] Baran O, Aykac A. The effect of fear of covid-19 transmission on male sexual behaviour: A cross-sectional survey study. Int J Clin Pract. 2021 Apr;75(4):e13889. doi: 10.1111/ijcp.13889. Epub 2020 Dec 12. PMID 33280187